## **Prespecified Analyses**

## 1) Effect of successful reperfusion in patients with anterior circulation strokes and large infarct core

<u>Population:</u> ASPECTS ≤5, anterior circulation LVO (intracranial ICA, Carotid-T, M1, M2)

Primary Outcome: mRS 0-3

Secondary Outcome: mRS 0-2

Safety Outcome: 3-month mortality, sICH

<u>Analysis:</u> Univariate comparison of outcome parameters in patients with and without successful reperfusion. Calculation of adjusted Odds Ratio of successful reperfusion (Thrombolysis in Cerebral Infarction 2b/3) for the primary and secondary outcomes with multivariable logistic regression adjusting for the following baseline confounders:

- Age (continuous)
- Sex (categorical)
- NIHSS admission (ordinal, per point increase)
- Tandem vs. non-Tandem (categorical, Tandem defined as >90% cervical stenosis or cervical occlusion)
- Center (contrast type: indicator, comparator: larges center, categorical)
- Risk Factor Hypertension (categorical)
- ASPECTS ≤3 vs ASPECTS 4-5 (categorical)
- IVT Bridging (categorical)
- Factor Dyslipidemia (categorical)
- Risk Factor Smoking (categorical)
- Risk Factors Previous Stroke (categorical)
- Risk Factor Diabetes (categorical)
- In Hospital Stroke (categorical)
- Type of Admission Imaging (CT vs MRI, categorical)
- Intracranial ICA/Carotid T vs M1/M2 (categorical)

<u>Additional Safety Analysis:</u> Comparison of sICH and interventional complications (classified as severe vasospasm, dissection, perforation and 'other') in patients with ASPECTS≤5 and ASPECTS 6-10.

Additional Sensitivity Analysis: Rerun logistic regression analysis with

- Confinement to ASPECTS ≤4,
- Add variable interaction term of successful reperfusion and admission modality
- Add interaction term for successful reperfusion and patients aged ≤70 years and >70 years.